CLINICAL TRIAL: NCT00411684
Title: A Prospective, Open-Label, Single Arm, Multicenter Study to Evaluate the Efficacy, Safety and Tolerability of CDB-2914 as Emergency Contraception When Taken Between 48 Hours and 120 Hours of Unprotected Sex
Brief Title: Safety and Efficacy of CDB-2914 for Emergency Contraception
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: HRA Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2914-005
Record Dates: First submitted 2006-12-13; First posted 2006-12-14 (Estimated); Results first posted 2021-05-03 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-04

CONDITIONS: Emergency Contraception
MeSH Terms: interventions — ulipristal

ARMS (1):
- CDB-2914 (Experimental): A Prospective, Open-Label, Single Arm, Multicenter Study to Evaluate the Efficacy, Safety and Tolerability of CBD-2914 as Emergency Contraception When Taken Between 48 Hours and 120 Hours of Unprotected Intercourse
  Interventions: Drug: CDB-2914

INTERVENTIONS:
Drug: CDB-2914

SUMMARY:
The purpose of this study is to assess the safety and efficacy of CDB-2914 for preventing pregnancy when taken 3 to 5 days after unprotected sexual intercourse.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or more
* Menstruating women with regular menstrual cycle between 24 and 35 days and intra-individual variations less than or equal to 5 days
* Request emergency contraception between 48 hours and 120 hours after unprotected intercourse as defined by lack of contraceptive use, or condom breakage (including condoms lubricated with spermicide) or other barrier contraceptive method failure
* No current use of hormonal contraception and having had at least one complete menstrual cycle (2 menses) since having stopped hormonal contraception
* For women with a recent history of Depo Provera use, the most recent injection must have been at least 9 months before study entry and followed by at least one complete menstrual cycle (2 menses)
* Willing to not use hormonal methods of contraception until study completion
* At least one complete menstrual cycle (2 menses) post delivery, miscarriage or abortion
* Able to provide informed consent in English
* Give voluntary, written informed consent, and agree to observe all study requirements (the subject needs to be available for follow-up over the next 6 weeks)
* Willing to abstain from further acts of unprotected intercourse during participation in the study and until pregnancy status has been ascertained

Exclusion Criteria:

* One or more acts of one unprotected intercourse more than 120 hours before requesting emergency contraception in the current cycle
* All acts of unprotected intercourse (in the current cycle) within 48 hours of presentation
* Currently pregnant as confirmed by positive HSUP test performed at screening
* Currently breast-feeding
* Current use of hormonal contraception
* Use of hormonal emergency contraception since last menstrual period
* Current use of IUD
* Tubal ligation
* Partner with a vasectomy
* Unsure about the date of the last menstrual period
* Severe asthma insufficiently controlled by oral glucocorticoid
* Currently enrolled in any other trial of an investigational medicine

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1623 (Actual)
Dates: Start 2006-11; Primary Completion 2008-04-08 (Actual); Study Completion 2009-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Fine, MD, Principal Investigator — Planned Parenthood of Houston and Southeast Texas
Locations (17):
- United States (17):
  - Planned Parenthood of Mar Monte, San Jose, California
  - Planned Parenthood of the Rocky Mountains, Denver, Colorado
  - Planned Parenthood of Greater Miami, Palm Beach and Treasure Cost, Miami, Florida
  - Planned Parenthood of South Palm Beach, Pembroke Pines, Pembroke Pines, Florida
  - Planned Parenthood of Indiana, Bloomington, Indiana
  - Planned Parenthood of Greater Iowa, Ames, Iowa
  - Planned Parenthood of Maryland, Baltimore, Maryland
  - Planned Parenthood League of Massachusetts, Boston, Massachusetts
  - Planned Parenthood of Mid-Michigan Alliance, Ann Arbor, Michigan
  - Planned Parenthood of Minnesota, Minneapolis, Minnesota
  - Planned Parenthood of Greater Cleveland, Cleveland, Ohio
  - Planned Parenthood of Columbia-Willamette, Portland, Oregon
  - Planned Parenthood of SE Philadelphia, Philadelphia, Pennsylvania
  - Planned Parenthood of the Texas Capital Region, Austin, Texas
  - Planned Parenthood of Houston and Southeast Texas, Houston, Texas
  - Planned Parenthood Association of Utah, Salt Lake City, Utah
  - Planned Parenthood of Western Washington, Seattle, Washington

REFERENCES:
- [Result] Fine P, Mathe H, Ginde S, Cullins V, Morfesis J, Gainer E. Ulipristal acetate taken 48-120 hours after intercourse for emergency contraception. Obstet Gynecol. 2010 Feb;115(2 Pt 1):257-263. doi: 10.1097/AOG.0b013e3181c8e2aa. PMID 20093897

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Screening 1623 Screening failures 90 Enrolled 1533
Groups:
- CDB-2914: A Prospective, Open-Label, Single Arm, Multicenter Study to Evaluate the Efficacy, Safety and Tolerability of CBD-2914 as Emergency Contraception When Taken Between 48 Hours and 120 Hours of Unprotected Intercourse
  CDB-2914
Period: Overall Study
Arm/Group | CDB-2914
Started | 1533
Completed | 1241
Not Completed | 292

BASELINE CHARACTERISTICS:
Population: ITT population
Groups:
- Exp Arm: A Prospective, Open-Label, Single Arm, Multicenter Study to Evaluate the Efficacy, Safety and Tolerability of CBD-2914 as Emergency Contraception When Taken Between 48 Hours and 120 Hours of Unprotected Intercourse
  CDB-2914
Arm/Group | Exp Arm
Number analyzed (Participants) | 1533
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1533
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.4 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1533
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 338
  Not Hispanic or Latino | 1182
  Unknown or Not Reported | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 21
  Asian | 35
  Native Hawaiian or Other Pacific Islander | 11
  Black or African American | 328
  White | 921
  More than one race | 212
  Unknown or Not Reported | 5
Region of Enrollment [Number; unit: participants]
  United States | 1533

OUTCOME MEASURES:

1. Primary Outcome: Pregnancy Rate
Description: A high sensitivity pregnancy test was performed at inclusion (between 48h and 120h after unprotected intercourse) and then until menses occured or up to 60 days if they did not, at the following time points:
  * 5-7 days after expected date of menses
  * 1 week later
  * every two week after
Time Frame: Up to 60 days after enrollment
Population: Primary efficacy population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CDB-2914
Number analyzed (Participants) | 1241
percentage of participants | 2.1 [1.4 to 3.1]

2. Secondary Outcome: Prevented Fraction (Number of Prevented Pregnancies Divided by the Number of Expected Pregnancies)
Description: Number of prevented pregnancies divided by the number of expected pregnancies
Time Frame: within the menstrual cycle of the unprotected Intercourse
Population: Primary efficacy population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CDB-2914
Number analyzed (Participants) | 1241
percentage of participants | 62.3 [41.9 to 75.6]

3. Secondary Outcome: Impact on Menstrual Bleeding Patterns
Description: Menstrual cycle length post treatment
Time Frame: within the menstrual cycle of the unprotected Intercourse
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | CDB-2914
Number analyzed (Participants) | 1533
Days | 31.8 (10.2)

4. Secondary Outcome: Frequencies of Subjects With Treatment Emergent Adverse Events
Description: Most common related adverse events in ITT population.
Time Frame: 12-14 days after expected menses
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | CDB-2914
Number analyzed (Participants) | 1533
percentage of participants
  Headache | 9.3
  Nausea | 9.2
  Abdominal pain | 6.8
  Dysmenorrhea | 4.1
  Dizziness | 3.5
  Fatigue | 3.4

ADVERSE EVENTS:
Arm/Group | CDB-2914
Serious Adverse Events (participants affected / at risk) | 1/1533
Other Adverse Events (participants affected / at risk) | 557/1533
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CDB-2914 (N=1533)
Seizure (Nervous system disorders) | 1 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CDB-2914 (N=1533)
Headache (Nervous system disorders) | 143 (143)
Nausea (Gastrointestinal disorders) | 141 (141)
Abdominal pain (Gastrointestinal disorders) | 104 (104)
Dysmenorrhea (Reproductive system and breast disorders) | 63 (63)
Dizziness (Nervous system disorders) | 54 (54)
Fatigue (General disorders) | 52 (52)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No